CLINICAL TRIAL: NCT00678782
Title: Evaluation of The Efficacy And Safety of Intra-Articular Etanercept in Patients With Refractory Knee Joint Synovitis: a Placebo Controlled, Single-Blind, Crossover-Trial, With Randomisation of Treatment Sequence
Brief Title: Evaluation of The Efficacy And Safety of Intra-Articular Etanercept in Patients With Refractory Knee Joint Synovitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Padova (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry); Azienda Ospedaliera di Padova (Other)
Responsible Party: Prof. Ugo Fiocco, Centro Multidisciplinare di Day Surgery, Azienda Ospedaliera di Padova
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: E-IA-02
Record Dates: First submitted 2008-05-14; First posted 2008-05-16 (Estimated); Last update posted 2008-05-16 (Estimated); Status verified 2008-05

CONDITIONS: Persistent Knee Joint Synovitis
Keywords: knee; synovitis; arthritis; rheumatoid arthritis; psoriatic arthritis; spondyloarthropathies; intraarticular; etanercept
MeSH Terms: conditions — Synovitis; Arthritis; Arthritis, Rheumatoid; Arthritis, Psoriatic; Spondylarthropathies | interventions — Etanercept

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: etanercept — etanercept 12.5mg, intraarticular injection administered once every two weeks for an eight week period
  Other Names: Enbrel
Drug: placebo — Placebo (NaCl) 0.5 ml intraarticular injection
  Other Names: NaCl

SUMMARY:
To assess the therapeutic efficacy, of the clinical response of intraarticular (IA) etanercept (E) 12.5 mg or placebo (P: NaCl) injections into single knee arthritic joint of patients with refractory knee joint synovitis (KJS), administered once every two week, for eight weeks, with cross over after 2 weeks, in two groups of randomly assigned patients, for whom traditional systemic disease-modifying antirheumatic drugs (DMARDs) is insufficient or inappropriate. The primary outcome measure is the Thompson articular index of KJS disease activity.

DETAILED DESCRIPTION:
The study is a single centre, placebo-controlled, single-blind, cross-over trial, with randomization of treatment sequence and open-label extension to be conducted in rheumatoid arthritis, psoriatic arthritis and spondyloarthropathies patients with resistant knee joint synovitis (KJS).

Patients are eligible if they suffered from persistent active KJS (characterized by pain, tenderness, and effusion), which had proved resistant to surgical treatment or to repeated IA corticosteroid therapy, or unresponsive to a minimum of 6 months second-line drug therapy with DMARD-, and/or anti-TNFα biologic agent monotherapy and systemic oral corticosteroid treatment, or to a combination therapy (drug failure is defined as discontinuation because of intolerable adverse effects or lack of clinical efficacy).

Concomitant Treatments: stable, appropriate doses of DMARDs (methotrexate, sulfasalazine, hydroxychloroquine, cyclosporine), DMARD combinations or low dose oral corticosteroids (≤10 mg prednisone) with or without non-steroid anti-inflammatory agents will be continued throughout the study.

Patients will be permitted stable doses (no greater than the maximum dose recommended by the manufacturer) of non-steroidal anti-inflammatory drugs (NSAIDs) but will be permitted to use only one NSAID at any given time. No analgesic could be taken before undergoing assessment on the day clinical evaluations will be performed.

Treatment: Each dose of study drug will be administered as one intraarticular (IA)injection carried out in each single knee joint that will be randomly assigned to blind treatment with 0.5 ml of etanercept (E) (12.5mg) or placebo (P) (NaCl). The IA injection will be administered once every two weeks for an eight week period. After 2 weeks time the patients will be crossed-over and each arthritic knee joint will receive E (12.5 mg) for four times or P for three times, respectively, administered every two weeks for an eight week period. All the IA injections will be administered after synovial fluid aspiration by the same operator. The study, patients with KJS flare up after IA injection will be asked to enter the open-label IA extension treatment with IA-E injection once every two weeks, for eight weeks.

Safety assessment: routine chemistry, haematology and urinalysis assessments will be performed at the screening, baseline and final examinations. Tuberculosis screening will be performed at the onset of the study. Patients will be evaluated clinically for adverse events at each examination. Local tolerance at the injection site(s) will be evaluated at all the controls.

Assessment of the patients' response: will be performed at baseline (T0) and at 2 (T2), 4 (T4), 6 (T6), and 8 (T8) weeks, and at the end of the 10 week single-blind, cross-over study or at the end of the open-label IA extension-study (up to 14 weeks) (Tend).

The primary efficacy endpoint is the Thompson articular index (THOMP) sum of scores for each knee joint, of pain on movement (0-3), soft tissue swelling (0-3) and warmth (0-3); (range 0-9). Secondary endpoints are: the Knee joint articular index (KJAI): the sum of the tenderness scores (0-3), joint swelling (0-3), the ballottement of patella or the "bulge sign" (0-2), and range of knee joint flexion (0-3) and extension (0-3) (KJAI, range 0-14). Standard joint evaluation comprise: the 66/68 swollen joint number (SJN) and tender joint number (TJN) (0-1); a modified Ritchie articular index (RAI), by assessment of 30 joints for tenderness (0-3) (range: 0-90), (including hand and foot distal interphalangeal joints (DIP) of each side as a group; the pain visual analogue scale (VAS) (0-100mm), the health assessment questionnaire (HAQ)- disability index (0-3) and the SF36 (range 0-24) at the above time points.

The serum CRP, the ESR, and the maximal synovial thickness (measured by grey-scale ultrasonography and contrast-enhanced magnetic resonance imaging) will be assessed at baseline and at the end of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18 years of age or older and of legal age of consent.
* A negative serum pregnancy test at screening and use of a medically acceptable form of contraception starting at screening and continuing throughout the study, is required for all females of childbearing potential (defined as an oral, injectable, or implantable contraceptive, intrauterine device, or barrier method combined with a spermicide).
* Meet the 1987 American Rheumatism Association (ARA) revised criteria for Rheumatoid Arthritis(RA) and generally accepted criteria for psoriatic (PsA) or spondyloarthritides (SpA).
* Meet the following criteria at both the screening visit and the baseline visit:

  * Refractory KJS defined by the presence of: Persistence of active synovitis of the knee (characterized by pain, tenderness and effusion), which had proved resistant to at least 6 months second-line DMARD therapy
  * Failure drug therapy with at least one DMARD and/or anti-TNFα biologic agent, and/or systemic or IA corticosteroid treatment. (Drug failure is defined as a drug discontinuation because of lack of clinical efficacy or intolerable adverse effects).
* Normal chest X-ray as clinically indicated.
* Provide written informed consent.
* In the opinion of the investigator, the patient will be able to comply with the requirements of the protocol.

Exclusion Criteria:

* Uncooperative patients with a history of poor compliance.
* Known hypersensitivity to etanercept or any of its components.
* Known significant concurrent medical disease including:

  * cancer or history of cancer (other than resected basal cell carcinoma of the skin)
  * congestive heart failure
  * myocardial infarction within 12 months of the screening visit
  * uncontrolled angina pectoris
  * active infection
  * sepsis or at risk of sepsis
  * severe pulmonary disease
  * known HIV infection
  * liver function abnormality (SGOT/AST, SGPT/ALT: greater than two times the upper limit of normal); liver cirrhosis or fibrosis
  * renal disease (creatinine level >175umol/L)
  * leukopenia (white blood cells <3.5 x 109/L)
  * thrombocytopenia (<1.25 x 1011/L)
  * haemoglobin </= 8.5 g/dL
* Females who are pregnant, breast feeding or at risk of pregnancy and not using a medically acceptable form of contraception.
* Any condition judged by the investigator that would cause the study to be detrimental to the patient.
* Use of any investigational drug within four weeks of the screening visit.
* In the opinion of the investigator, the patient shows persistent signs of immunosuppression.
* Receipt of any live attenuated vaccine within eight weeks before the screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2005-04; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Thompson articular index | 2 weeks

SECONDARY OUTCOMES:
Knee Joint Articular Index | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ugo Fiocco, MD, PhD, Principal Investigator — University of Padova
Locations (1):
- Centro Multidisciplinare di Day Surgery, Azienda Ospedaliera di Padova, Ospedale Busonera, via Gattamelata 64, Padua, Italy

REFERENCES:
- [Derived] Fiocco U, Sfriso P, Oliviero F, Lunardi F, Calabrese F, Scagliori E, Cozzi L, Di Maggio A, Nardacchione R, Molena B, Felicetti M, Gazzola K, Stramare R, Rubaltelli L, Accordi B, Costa L, Roux-Lombard P, Punzi L, Dayer JM. Blockade of intra-articular TNF in peripheral spondyloarthritis: its relevance to clinical scores, quantitative imaging and synovial fluid and synovial tissue biomarkers. Joint Bone Spine. 2013 Mar;80(2):165-70. doi: 10.1016/j.jbspin.2012.06.016. Epub 2012 Aug 3. PMID 22867975
- [Derived] Fiocco U, Oliviero F, Sfriso P, Calabrese F, Lunardi F, Scagliori E, Rubaltelli L, Stramare R, Di Maggio A, Nardacchione R, Cozzi L, Molena B, Felicetti M, Gazzola K, Lo Nigro A, Accordi B, Roux-Lombard P, Dayer JM, Punzi L. Synovial biomarkers in psoriatic arthritis. J Rheumatol Suppl. 2012 Jul;89:61-4. doi: 10.3899/jrheum.120246. PMID 22751595